CLINICAL TRIAL: NCT04042662
Title: Predictors and Outcomes of Meropenem Treatment Failure Among Patients With Septic Shock in Intensive Care Unit
Acronym: Meropenem
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Dr Mohd Zulfakar Mazlan, Research Supervisor, Universiti Sains Malaysia
Other Study IDs: MeropenemUSM
Record Dates: First submitted 2019-07-30; First posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-08

CONDITIONS: Predictors and Outcomes of Meropenem Treatment Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Meropenem Failure ( Treatment failure)
  Interventions: Other: no intervention
- Meropenem Success ( Treatment Success)
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Lately, the inappropriate used of Meropenem in critically ill patient were increased. Therefore, increased development of drug resistance bacteria towards Meropenem.

As known that Carbapenem-Resistance Enterobacteriaceae (CRE) is part of complication when Meropenem is widely used in the intensive care unit. CRE are very difficult to treat within Gram negative bacteria as it encodes Carbapenemase enzyme which breaks down Carbapenem anti-microbial such as Meropenem. The widespread carbapenemase production in the Enterobacteriaceae was unknown until the early 2000 until first reported in 2001. Despite that, most doctors and physician favourite, and still prescribe Meropenem as the antibiotic of choice for the critically ill patients empirically. This is because of its broad spectrum of coverage for bacteria. Thus, a number of Meropenem treatment failure were increased as resistance increase.This study will evaluate the appropriate use of Meropenem and determine the predictors of Meropenem treatment failure as well as the patient outcomes.As a result, it can be a guidance prior prescribing the Meropenem base on patient clinical condition and parameters while balancing the risk and benefits of its used.

ELIGIBILITY:
Inclusion Criteria:

1. Septic shock patient admitted to ICU
2. Age equal or more than 18 years old (No upper limit of age)
3. Receive Meropenem for at least 3 days

Exclusion Criteria:

1. Meropenem as prophylaxis
2. Patient who had culture Carbapenem Resistant Enterobacteriaceae organism (CRE)
3. Patient who admitted with proven diagnosis of Cardiogenic shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Reference population is septic shock patient who was prescribed with Meropenem and admitted to ICU HUSM from 01/01/2016 - 01/06/2019
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-08-05 (Estimated); Primary Completion 2020-08-05 (Estimated); Study Completion 2020-08-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment failure with antibiotic meropenem as assessed by clinical criteria of sepsis parameters among patient | 3 years
  with septic shock in intensive care unit.
Number of factors associated with antibiotic meropenem treatment failure among patient | 3 years
  with septic shock in intensive care unit.
Number of the patients who die after treated with antibiotic meropenem in intensive care unit | 3 years
  Mortality

IPD SHARING:
Plan to Share IPD: No